CLINICAL TRIAL: NCT04161586
Title: Prilocaine for Spinal Anesthesia in Ambulatory Setting: an Observational Retrospective Study
Brief Title: Prilocaine for Spinal Anesthesia in Ambulatory Setting
Status: Completed | Type: Observational
Sponsor: Ospedale di Circolo - Fondazione Macchi (Other)
Responsible Party: Principal Investigator, Andrea Luigi Ambrosoli, Anesthesia and Intensive Care Chief - Ospedale Filippo Del Ponte, Ospedale di Circolo - Fondazione Macchi
Other Study IDs: VAR-005
Record Dates: First submitted 2019-11-09; First posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Anesthesia, Spinal; Prilocaine; Ambulatory Surgical Procedures
Keywords: Spinal Anesthesia; Prilocaine; Ambulatory Surgery; Safety
MeSH Terms: interventions — Prilocaine; Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Prilocaine Hydrochloride — Spinal Prilocaine for Ambulatory Surgery
  Other Names: Spinal Anesthesia

SUMMARY:
The purpose of this study is to retrospectively analyze data from more than 3000 procedures, to better define the safety profile of spinal prilocaine and the incidence of complications and side effects.

DETAILED DESCRIPTION:
We designed a retrospective cohort study to analyze the safety profile and the incidence of side effects associated with prilocaine for spinal anesthesia in ambulatory settings.

Data will be obtained from an internal database where are prospectively recorded clinical data from spinal anesthesia consecutively performed with prilocaine at our institution for ambulatory surgery from 2011 to 2019. Variables recorded in the database and analyzed will include demographic data, type of surgery, presence of surgical, anesthesiological or general complications, need for unplanned admission and percentage of completed database records.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory surgical procedures performed under spinal anesthesia with Prilocaine

Exclusion Criteria:

* General Anesthesia
* Procedures lasting longer than 2 hours

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Single Center Ambulatory Surgical Patients
Sampling Method: Non-Probability Sample
Enrollment: 3291 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-11-09 (Actual)

PRIMARY OUTCOMES:
anesthesia-related complication | 2011-2019
  urinary retention, lipotimia, postoperative nausea, arrhythmia, hypotension, transient neurological symptoms, headache

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Day Surgery Ospedale di Circolo Varese, Varese, VA, Italy